CLINICAL TRIAL: NCT02855255
Title: Comparing the 26 Week Efficacy of Allen Carr's Easyway to Stop Smoking and NHS 1-1 Counselling Provision
Brief Title: Study Comparing Two Stop Smoking Intervention Efficacies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London South Bank University (Other)
Collaborators: NHS Lambeth (Other); NHS Southwark CCG (Other); Allen Carr Easyway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 7697
Record Dates: First submitted 2016-07-07; First posted 2016-08-04 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NHS smoking cessation (Active Comparator): NHS 1-1 smoking cessation programme. One thirty minute session followed by up to five shorter sessions (approx.10/15minutes) comprising Cognitive Behavioural Therapy/Motivational Interviewing to assist with smoking cessation.
  Interventions: Behavioral: NHS 1-1 smoking cessation programme.
- Allen Carr's Easyway smoking cessation (Active Comparator): Group smoking cessation programme. One 5/6 hour group session (plus one or two 3 hour booster sessions over the following 3 months for those who require them) comprising of Allen Carr's Easyway method being delivered in a spoken form.
  Interventions: Behavioral: Group smoking cessation programme

INTERVENTIONS:
Behavioral: NHS 1-1 smoking cessation programme. — Smoking cessation using cognitive behavioural therapy/motivational interviewing
  Arms: NHS smoking cessation
Behavioral: Group smoking cessation programme — Smoking cessation using Allen Carr's Easyway method being delivered in a spoken form.
  Arms: Allen Carr's Easyway smoking cessation

SUMMARY:
The proposed study will compare the efficacy of two psychological stop smoking interventions.

DETAILED DESCRIPTION:
The proposed study comprises a randomised controlled trial (n = 620) which will compare the efficacy of two psychological stop smoking interventions. Specifically, Allen Carr's Easyway smoking cessation programme comprising one 5/6 hour group session (plus one or two 3 hour booster sessions over the following 3 months for those who require them) and a 1-1 counselling service available via the NHS (comprising one 30 minute session and four weekly follow ups of 10-15 minutes) will be compared. The efficacy of both treatments will be followed up at 4, 12 and 26 weeks after treatment. The evaluation will be compliant with the Russell 6 Standard (which requires, amongst other things, a double blind, randomised design, chemical verification of quit outcomes, and the inclusion of all participants who received treatment in the final analysis). The findings will add to the evidence base around the use of the Allen Carr method, in particular by testing it in non-commercial settings.

ELIGIBILITY:
Inclusion Criteria:

Current smoker Aged over 18 Prepared to be assigned randomly to one of two treatment conditions (NHS standard provision or Allen Carr's Easyway) Intend to quit smoking cigarettes.

Exclusion Criteria:

Individuals who would prefer an NHS provided treatment Currently in another RCT or similar research project Have a mental health condition Are pregnant Have a respiratory disease (such as chronic obstructive pulmonary disease or emphysema).

Unable to reach the treatment locations (London South Bank Universities Southwark Campus or SW20) .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 620 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-05-25 (Actual)

PRIMARY OUTCOMES:
Cessation of smoking | 26 weeks post treatment commencement
  Measured in line with the Russell 6 standard (i.e. fewer than 5 incidents of smoking from the quit date, including all participants lost to follow-up as failed treatment, and confirming all successful quits via breath carbon monoxide testing). The intention to treat principle will be followed, and those lost to follow-up will be considered failed quit.

SECONDARY OUTCOMES:
Self-reported maintenance of smoking cessation questions | 4, 12, 26 weeks post treatment commencement
  current cessation, number of slips, number of cigarettes in past week/month/since last session.
The Satisfaction with Life Scale (Diener, Emmons, Larsen, & Griffin, 1985). | Baseline and 4, 12, 26 weeks post treatment commencement
  A 5-item scale designed to measure global cognitive judgements of one's life satisfaction. Participants indicate how much they agree or disagree with each of the 5-items using a 7-point scale that ranges from 7 Strongly agree to 1 Strongly disagree.
Survey assessing use of Nicotine replacement therapy/nicotine containing products | 4, 12, 26 weeks post treatment commencement
  Participants will be asked to answer Yes/No to the following: 'Since we last met, have you regularly used any of the following?' and 'Are you planning on using any of the following in the future?' E-cigarettes, Nicotine Patches, Nicotine Gum, Other.
Quit efficacy questionnaire | Baseline, 4, 12, 26 weeks post treatment commencement
  Measured on a scale of 1-7 (strongly disagree - strongly agree), to the following items: 'I can achieve my aims to quit smoking', 'I can cope with the demands of quitting smoking', 'It is unlikely that I will do well at quitting smoking', 'I think I can perform well at quitting smoking'.
Perceived value of being nicotine free - Questionnaire | 4, 12, 26 weeks post treatment commencement
  Measured on a scale of 1-7 (strongly disagree - strongly agree), to the following items: 'Being nicotine free is of value to me', 'I value being nicotine free', 'Having no nicotine in my system is / would be beneficial to me'.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Frings, PhD, Principal Investigator — London South Bank University
Locations (1):
- London South Bank University, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared at participant by participant level in an anonymous form via it being lodged with an appropriate data repository, alongside London South Bank University's own repository.

REFERENCES:
- [Derived] Wood KV, Albery IP, Moss AC, White S, Frings D. Study protocol for a randomised controlled trial of Allen Carr's Easyway programme versus Lambeth and Southwark NHS for smoking cessation. BMJ Open. 2017 Dec 14;7(12):e016867. doi: 10.1136/bmjopen-2017-016867. PMID 29247083